

### Anexo 6. F-06 Consentimiento Informado para pacientes

Es probable que el presente formulario de consentimiento contenga palabras o conceptos que usted no entienda. Por favor, pídale al investigador o a los asistentes del estudio que le expliquen todas las palabras, conceptos o información que no comprenda con claridad. Igualmente, puede realizar todas las preguntas que considere sean necesarias para tomar la decisión, tómese el tiempo necesario para pensar y, si es del caso, consulte a familiares, amigos o personas allegadas que le ayuden a comprender mejor las razones para aceptar su inclusión en la investigación.

## Investigadores:

Juan Diego Lemos Duque (Investigador principal)
Juan Guillermo Barreneche (Coinvestigador)
Sofía Catalina Henao Aguirre (Coinvestigadora)
Ana María Posada (Coinvestigadora)
Sara Salazar Salgado (Coinvestigadora)
Jenny Kateryne Aristizabal Nieto (Coinvestigadora)
Juan Gabriel Arboleda Ramírez (Coinvestigador)
Maria Bernarda Salazar Sánchez (Coinvestigadora)

Rehabilitación en Salud de la Universidad de Antioquia.

| 1. Introduccion | | | | |
|---|---|---|---|---|
| A usted Señor(a) | | <b>,</b> | identificada | con |
| documento de identidad | de | , se le está invitando a partic | ipar en un est | udio |
| de investigación de los grupos d | e Bioinstrumentación | e Ingeniería de Rehabilitación – GIBI | C v del Grupe | o de |

En primer lugar, usted debe conocer que la participación en el estudio es absolutamente voluntaria. Esto quiere decir que si usted lo desea puede negarse a participar o retirarse del estudio en cualquier momento sin tener que dar explicaciones. En caso de que desee participar, se le entregara copia diligenciada y firmada del consentimiento informado.

Sitio donde se llevará a cabo el estudio: Prótesis Avanzadas S.A.S. Entidad que respalda la investigación: Universidad de Antioquia Entidades que patrocinan la investigación:

- \*Minciencias
- \*Universidad de Antioquia
- \*Prótesis avanzadas S.A.S.

# 2. Información sobre el estudio.

# Propósito

Para las personas que han tenido una amputación de miembro superior, un aspecto de su rehabilitación es usar una prótesis que les permita recuperar una parte de la función perdida, permitiéndoles ganar autonomía y mejorar su calidad de vida. En un país como Colombia el acceso a estos dispositivos costosos fabricados en otros países es difícil. Esto último hace que, en nuestro país, la mayoría de la población no tenga acceso a este tipo de tecnologías y, por tanto, se les dificulte trabajar, estudiar y desempeñar otras actividades que les permitan mejorar su calidad de vida.



El objetivo principal de este estudio es diseñar, implementar y evaluar la efectividad de una prótesis mioeléctrica que permita la rehabilitación física de personas con amputación transrradial (A nivel del antebrazo).

Es importante aclarar que el resultado final de este proyecto será el diseño de una prótesis mioeléctrica. La metodología se dividirá en varias fases para la definición de los objetivos que se esperan satisfacer con el diseño de las prótesis hasta la creación de un prototipo funcional y la realización de pruebas con personas como usted.

#### **Procedimientos**

Todos los pacientes (Doce en total) serán evaluados por un médico fisiatra o una terapeuta quienes verificarán si cumple con los criterios para ingresar al estudio.

Una vez elegidos, los pacientes participarán en dos fases:

<u>+Diseño conceptual:</u> En una sesión presencial (Individual o grupal) se evaluarán las prioridades y preferencias de los pacientes con respecto al uso de prótesis y a las necesidades que éstas deberían cubrir. Se indagará por aspectos como la usabilidad, el confort, la adaptación, la fuerza, la movilidad, el desempeño en las actividades de la vida diaria y la calidad de vida. Adicionalmente, para definir el diseño de la prótesis se obtendrán datos de los pacientes acerca del funcionamiento (Movilidad, fuerza, precisión en agarres) y se tomarán moldes y medidas para la elaboración de la prótesis.

<u>+Evaluación de efectividad:</u> Luego de definir los aspectos conceptuales se diseñará y elaborará una prótesis mioeléctrica. Cada prótesis será entregada por integrantes del equipo de diseño y un terapeuta físico u ocupacional, quienes entrenarán en el uso de ésta y realizarán los ajustes necesarios para su adaptación en dos sesiones de 3 horas cada una.

Para demostrar la efectividad de la prótesis se utilizarán cuestionarios de funcionamiento (desempeño en actividades de la vida diaria), satisfacción con la prótesis y calidad de vida relacionada con la salud y además se realizarán pruebas de desempeño con y sin la prótesis, bajo observación por uno de los investigadores. Esto se realizará en dos momentos para evaluar las diferencias con y sin el uso de prótesis. Todos los pacientes recibirán la prótesis y se asignará de manera aleatoria (al azar) el momento para su uso. En total se tienen programadas dos mediciones, es decir, momentos de evaluación.

# Inconvenientes, malestares y riesgos

Los procedimientos realizados son considerados de bajo riesgo. En cada paciente se evaluarán aspectos clínicos (Movilidad, fuerza, precisión en agarres) y del funcionamiento mediante pruebas físicas. Además, se aplicarán cuestionarios para recoger datos sobre el desempeño en las actividades de la vida diaria, la satisfacción con la prótesis y la calidad de vida. También se tomarán moldes y medidas para la elaboración de la prótesis, lo cual no ocasionará malestar físico ni riesgo para el paciente. Esto implicará desplazamientos al sitio designado para tal fin, cuyos costos serán asumidos por los investigadores.

En el momento de entrega y adaptación de la prótesis se realizarán los ajustes necesarios para corregir cualquier causa de molestia relacionada con el uso de la prótesis. Los investigadores no se comprometen a realizar tratamientos ni asumir costos en el caso de complicaciones no relacionadas con el uso de la prótesis sino secundarias a la amputación o como consecuencia de la evolución natural de ésta (Por ejemplo: Dolor de miembro fantasma) o de otras no relacionadas con la amputación.

Cabe aclarar que las prótesis se clasifican como dispositivos médicos no son invasivos y que la empresa Prótesis Avanzadas cuenta con experiencia en la producción y adaptación de prótesis en impresión 3D para miembro superior.

El paciente no tendrá que asumir gastos adicionales que no estén previstos en el estudio.

#### Beneficios

Los participantes del estudio no recibirán ningún beneficio económico por participar en éste. La razón por la cual se le invita a participar es la contribución para el desarrollo de la ciencia y el entendimiento.



La información personal que usted dará a nuestros investigadores en el curso de este estudio permanecerá en secreto y no se proporcionará a ninguna persona diferente a usted, será custodiada por los investigadores formularios de encuestas serán archivados en una base de datos de la Universidad de Antioquia. Cuando haya concluido este estudio los participantes tendrán derecho a conocer los resultados de la investigación.

En caso de que se presente cualquier duda o pregunta sobre los procedimientos, inconvenientes, riesgos y beneficios de este estudio, serán resueltos por parte de cualquiera de los investigadores durante el tiempo del estudio.

En caso de que se presenten dudas por fuera de estos tiempos serán solucionadas por:

Juan Diego Lemos Duque Investigador del Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) E-mail: juan.lemos@udea.edu.co Teléfono: 219 8588

Facultad de Ingeniería Universidad de Antioquia

Gabriel Jaime Montoya Presidente Comité de Bioética E-mail: bioeticamedicina@udea.edu.co Teléfono: 2196065

Teléfono: 2196065 Facultad de Medicina

### 3. Información complementaria

Usted debe tener en cuenta los siguientes puntos en caso de decidir participar en esta Investigación.

# Derecho a retirarse del estudio de investigación.

Usted puede retirarse del estudio en cualquier momento, sin embargo, los datos obtenidos hasta ese momento seguirán formando parte del estudio a menos que usted solicite expresamente que su identificación y su información sea borrada de nuestra base de datos.

Adicionalmente su participación también terminará cuando el estudio haya concluido, lo cual está destinado para una duración de 24 meses.

#### Obligaciones del participante:

- 1) Asistir a los seguimientos y controles por equipo médico y de diseño.
- 2) Colaborar en el diligenciamiento de los cuestionarios y encuestas mencionadas.
- 3) Proporcionar una información fidedigna a los investigadores.

### Obligaciones del investigador.

- 1) Seguimiento del paciente.
- 2) Solución de los problemas que surjan de la investigación.
- 3) Conexión de los pacientes con los servicios médicos que se requieran.
- 4) Guardar la confidencialidad de los datos del participante.

#### **Resultados esperados**

Se espera conocer las preferencias, prioridades y objetivos de las prótesis que permitan mejorar el funcionamiento y desempeño de los pacientes en actividades de la vida diaria. Como producto final se espera diseñar y adaptar una prótesis mioeléctrica para amputación transrradial.



# 4. Consentimiento informado

Después de haber leído y comprendido el contenido de este documento con relación al estudio y habiendo dispuesto de tiempo suficiente para reflexionar sobre las implicaciones de mi decisión, libre, consciente y voluntariamente manifiesto que no he recibido presiones verbales, escritas y/o mímicas para participar en el estudio; que dicha decisión la tomó en pleno uso de mis facultades mentales, sin encontrarme bajo efectos de medicamentos, drogas o bebidas alcohólicas, consciente y libremente.

| medicamei | itos, urogas o bebluas a | ilcoriolicas, corisciei | ite y libremente. | |
|---|---|---|---|---|
| | encia, firmo este docun<br>, del mes de | | iento informado, en la ciudad de<br> | , el |
| Participant | e | | | |
| Nombre | | | _ | |
| CC | de | | | |
| Firma | | | | |
| Testigo 1 | | | | |
| Nombre | | | _ | |
| CC | de | | | |
| Parentesco | | | | |
| Testigo 2 | | | | |
| Nombre | | | _ | |
| CC | de | | | |
| Parentesco | | | | |